CLINICAL TRIAL: NCT07184853
Title: Prospective Multicenter Randomized Study of Ruxolitinib Plus Etanercept vs Ruxolitinib Alone for Corticosteroid-Refractory Severe Acute GVHD After Allogeneic HSCT
Brief Title: Ruxolitinib Plus Etanercept vs Ruxolitinib for Steroid-Refractory Severe Acute GVHD
Acronym: RESCUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yanmin Zhao, Vice Director, Bone Marrow Transplantation Center, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rux-Eta-SR-aGVHD
Record Dates: First submitted 2025-08-27; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Graft vs Host Disease
Keywords: Ruxolitinib; Etanercept; JAK1/2 inhibitor; TNF-α inhibitor; Corticosteroid-refractory GVHD; Severe aGVHD; Allo-HSCT complications; Graft-versus-Host Disease treatment; Immunosuppression
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib; Etanercept

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by GVHD grade (III vs IV) and then randomized in a 1:1 ratio to receive either ruxolitinib alone or ruxolitinib plus etanercept.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib Monotherapy (Active Comparator): Participants will receive ruxolitinib (10 mg orally twice daily, approximately every 12 hours, with or without food). Treatment will continue for up to 24 weeks. Dose reductions or discontinuation may occur according to protocol-defined safety and response criteria. Corticosteroid tapering will follow study guidelines.
  Interventions: Drug: Ruxolitinib (JAKAVI®)
- Ruxolitinib Plus Etanercept (Experimental): Participants will receive ruxolitinib (10 mg orally twice daily, approximately every 12 hours, with or without food) combined with etanercept (25 mg subcutaneous injection, twice weekly for 4 weeks, total 8 doses). Etanercept may be extended for an additional 2-4 weeks at investigator's discretion for patients with partial response. Treatment with ruxolitinib may continue for up to 24 weeks, with dose tapering per study protocol. Corticosteroid tapering will follow study guidelines.
  Interventions: Drug: Ruxolitinib (JAKAVI®); Drug: Etanercept (Enbrel)

INTERVENTIONS:
Drug: Ruxolitinib (JAKAVI®) — Ruxolitinib will be administered orally at a dose of 10 mg twice daily (approximately every 12 hours), with or without food. Dose modifications are allowed according to protocol-defined safety and efficacy criteria. Ruxolitinib may be continued for up to 24 weeks, with tapering guided by patient response and GVHD status.
Drug: Etanercept (Enbrel) — Etanercept will be administered as a subcutaneous injection at a dose of 25 mg twice weekly for 4 weeks (total 8 doses). For patients with partial response at day 28, treatment may be extended once weekly for an additional 2-4 weeks at the investigator's discretion.
  Arms: Ruxolitinib Plus Etanercept

SUMMARY:
This is a prospective, multicenter, randomized controlled trial designed to evaluate whether the combination of ruxolitinib and etanercept provides superior efficacy compared with ruxolitinib monotherapy in patients with severe corticosteroid-refractory acute graft-versus-host disease (SR-aGVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Acute graft-versus-host disease (aGVHD) is one of the most common and life-threatening complications following allo-HSCT. Although corticosteroids remain the standard first-line treatment, many patients do not respond adequately. For patients with severe steroid-refractory aGVHD, the prognosis is extremely poor, with high short-term mortality and very low long-term survival.

Ruxolitinib, a JAK1/2 inhibitor, has been approved for the treatment of SR-aGVHD, but response rates remain suboptimal, particularly in patients with gastrointestinal involvement. Etanercept, a tumor necrosis factor-alpha (TNF-α) inhibitor, has shown activity in GVHD by targeting inflammatory pathways. Previous observational studies from our center suggested that combining ruxolitinib with etanercept may improve response rates, especially in gastrointestinal and hepatic GVHD, without significantly increasing relapse risk.

In this trial, approximately 122 patients with grade III-IV SR-aGVHD will be randomized 1:1 to receive either ruxolitinib alone or ruxolitinib plus etanercept. The primary endpoint is the overall response rate (ORR) at day 28. Secondary endpoints include durable response, best overall response, failure-free survival, overall survival, cumulative incidence of relapse, non-relapse mortality, incidence of chronic GVHD, and safety outcomes.

This study seeks to provide new clinical evidence for an optimized treatment strategy for patients with severe SR-aGVHD, aiming to improve outcomes in this high-risk population.

DETAILED DESCRIPTION:
Steroid-refractory severe acute graft-versus-host disease (SR-aGVHD) remains a leading cause of early morbidity and mortality after allogeneic hematopoietic stem cell transplantation. Although ruxolitinib (JAK1/2 inhibition) improves outcomes versus best available therapy, non-response and limited durability-particularly with gastrointestinal involvement-underscore the need for rational combination strategies. Tumor necrosis factor-α (TNF-α) is a proximal driver of allo-inflammation; biomarker analyses suggesting elevated TNFR1 among non-responders to JAK inhibition support TNF-α pathway engagement as a potential mechanism of resistance. Prior single-arm, multicenter experience with ruxolitinib plus etanercept has shown encouraging activity in severe disease, including gastrointestinal and hepatic involvement, without an apparent increase in relapse risk, providing the rationale for this randomized evaluation.

This prospective, multicenter, randomized, open-label study tests whether adding etanercept to ruxolitinib improves clinical response at the prespecified primary assessment time point in patients with corticosteroid-refractory severe aGVHD after allogeneic transplantation. Participants are randomized 1:1 to combination therapy or ruxolitinib alone, with stratification by baseline disease severity to balance key prognostic factors across arms. The open-label design reflects practical differences in administration; where feasible, centralized or blinded review procedures are implemented to mitigate assessment bias.

Study treatment follows protocol-defined principles for initiation, modification, and discontinuation that align with current practice, including management algorithms for cytopenias, organ dysfunction, and relevant drug interactions. Systemic corticosteroids at enrollment are required for the SR definition; tapering after response is guided by predefined algorithms. Concomitant supportive care, infection prophylaxis, and transfusion support are provided according to institutional standards. Rescue therapy or treatment withdrawal is permitted under prespecified lack-of-benefit or safety criteria.

The primary objective is to determine superiority of combination therapy over ruxolitinib alone on clinical response at the primary time point. Key secondary objectives address response durability, transplant-related outcomes, corticosteroid exposure, and safety/tolerability; exploratory analyses include infection burden and biomarker assessments to characterize pharmacodynamic effects and response heterogeneity. Outcome definitions and time frames are specified in the Outcome Measures section; eligibility criteria are provided in the Eligibility section.

Safety is actively monitored throughout treatment and follow-up, with predefined surveillance for infections (including viral reactivation), cytopenias, and organ-specific toxicities. An independent safety review process periodically evaluates unblinded data per charter. The trial is sized to detect a clinically meaningful difference under conservative assumptions and includes longitudinal follow-up to capture durability, survival, and late safety signals, thereby informing whether dual pathway modulation (JAK and TNF-α) can improve outcomes in this high-risk population without unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Received allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source (matched sibling, matched unrelated, or haploidentical), using bone marrow, peripheral blood stem cells, or cord blood; conditioning regimen may be myeloablative, reduced-intensity, or non-myeloablative.

Age between 12 and 70 years.

Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.

Clinical diagnosis of grade III-IV acute graft-versus-host disease (aGVHD) according to MAGIC criteria.

Evidence of neutrophil and platelet engraftment prior to study treatment (absolute neutrophil count >1,000/mm³ and platelet count ≥20,000/mm³ within 48 hours before study entry; growth factor support and transfusion permitted).

Diagnosis of steroid-refractory aGVHD, defined as one of the following:

Disease progression after 3-5 days of methylprednisolone 2 mg/kg/day (or equivalent).

No improvement after 7 days of methylprednisolone 2 mg/kg/day (or equivalent).

Progression from grade II to grade III-IV aGVHD after 3-5 days of methylprednisolone 1 mg/kg/day (or equivalent).

Able to take oral medication.

Expected survival >8 weeks.

Women of childbearing potential must have a negative serum β-HCG test prior to enrollment; both male and female participants of reproductive potential must agree to use effective contraception during the study and for 3 months after study completion.

Voluntary written informed consent provided and ability to comply with study procedures.

Exclusion Criteria:

Prior systemic treatment for aGVHD other than corticosteroids with or without calcineurin inhibitors (CNI); prophylactic use of MTX, MMF, or CD25 monoclonal antibody is permitted.

Clinical features consistent with de novo chronic GVHD or overlap syndrome (per Jagasia 2015).

Uncontrolled active infection, including severe bacterial, fungal, viral, or parasitic infection. Patients on appropriate treatment without evidence of progression may be eligible.

Evidence of active tuberculosis.

Known HIV infection.

Relapse of primary malignancy or post-transplant lymphoproliferative disorder.

Severe respiratory disease, including mechanical ventilation or resting oxygen saturation <90%.

Renal dysfunction: serum creatinine >2.0 mg/dL, requirement for dialysis, or creatinine clearance <30 mL/min (Cockcroft-Gault).

Active hepatitis B infection (HBsAg positive with HBV DNA ≥1×10³ IU/mL) or active hepatitis C infection (HCV antibody positive with detectable HCV RNA above normal).

Clinically significant or uncontrolled cardiac disease, including recent myocardial infarction, uncontrolled hypertension, NYHA class III/IV heart failure, unstable angina, or clinically significant arrhythmia (e.g., sustained ventricular tachycardia, second- or third-degree AV block).

Cholestatic disease or unresolved hepatic veno-occlusive disease not attributed to aGVHD.

History of progressive multifocal leukoencephalopathy (PML).

Prior exposure to JAK inhibitors after allo-HSCT.

Participation in another investigational drug trial within 30 days or within 5 half-lives of the investigational drug (whichever is longer).

Prior history of grade ≥3 non-hematologic adverse events attributable to ruxolitinib or etanercept.

Any condition judged by the investigator to place the patient at undue risk or interfere with study participation.

Known hypersensitivity or intolerance to systemic immunosuppressive agents.

Pregnant or breastfeeding women.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Day 28 | From date of treatment initiation to Day 28.
  Proportion of patients achieving complete response (CR) or partial response (PR) compared with baseline organ staging, as assessed by MAGIC criteria.

SECONDARY OUTCOMES:
Durable Overall Response at Day 56 | From date of treatment initiation to Day 56.
  Proportion of patients who achieved a response at day 28 and maintained the same response at day 56.
Duration of Response (DOR) | From date of treatment initiation to the earliest of loss of response (per MAGIC criteria), initiation of new systemic therapy for aGVHD, or death; assessed up to 24 weeks after treatment initiation.
  From first documented response until progression of aGVHD or initiation of new systemic therapy for aGVHD, assessed up to 24 weeks
Best Overall Response (BOR) | From date of treatment initiation through Day 28.
  Proportion of patients achieving CR or PR at any time up to day 28, without requiring new systemic immunosuppressive therapy.
Failure-Free Survival (FFS) | From date of treatment initiation until event, assessed up to 24 weeks.
  Time from treatment initiation to relapse/progression of underlying hematologic disease, non-relapse mortality, or initiation of new systemic therapy for aGVHD.
Overall Survival (OS) | From date of treatment initiation until death, assessed up to 2 years.
  Time from treatment initiation until death from any cause.
Non-Relapse Mortality (NRM) | From date of treatment initiation until non-relapse death, assessed up to 2 years.
  Death without relapse or progression of underlying hematologic disease.
Cumulative Incidence of Relapse (CIR) | From date of treatment initiation until relapse/progression, assessed up to 2 years.
  Relapse or progression of the underlying hematologic disease.
Corticosteroid Use | From date of treatment initiation, assessed up to 24 weeks.
  Assessment of corticosteroid dose reduction and tapering patterns.
Incidence of Chronic GVHD | From date of treatment initiation, assessed up to 2 years.
  Cumulative incidence of chronic GVHD or overlap syndrome after study treatment.
Safety and Tolerability | From treatment initiation until 30 days after the end of study treatment.
  Incidence, severity, and duration of adverse events (AEs) and serious adverse events (SAEs), including infections and secondary malignancies, assessed according to CTCAE v5.0.

OTHER OUTCOMES:
Exploratory Biomarker Analyses | From date of treatment initiation, assessed up to 24 weeks.
  Evaluation of serum biomarkers (e.g., TNFR1) and other molecular correlates associated with response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No